CLINICAL TRIAL: NCT04576962
Title: County Level Correlates of HPV Vaccine Series Completion Among Children Ages 11-14 Years in Indiana
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gregory Zimet, Professor, Indiana University
Other Study IDs: MISP# 60560
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Human Papillomavirus Vaccination
Keywords: HPV Vaccines; Health Status; Access to Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 14 years or younger: All children in Indiana aged 14 years and younger who received the first dose of HPV vaccine during the 2017 and 2018 calendar years. This is a non-interventional study, with data to be analyzed at the county level only.
  Interventions: Other: Immunization Information System Review

INTERVENTIONS:
Other: Immunization Information System Review — Extraction of county- and state-level data on HPV vaccine completion from Indiana's Immunization Information System

SUMMARY:
The overall objective is to document geographic variability in HPV vaccine series completion across the state of Indiana and to identify factors associated with low versus high rates of completion.

Objective a: To map HPV vaccine series completion rates across Indiana's 92 counties for children aged 14 years and younger. Hypothesis: The investigators expect wide variability in completion rates from county to county. Further, the investigators expect significantly less variability in county-level administration of vaccines required for middle-school entry (Tdap, MenACWY, and HepA vaccines).

Objective b: To identify county-level characteristics associated with HPV vaccine series completion rates across Indiana's 92 counties. Hypothesis: The investigators expect factors reflective of pragmatic obstacles to be associated with lower completion rates: such as lower population density, fewer primary health care providers (HCP) per capita, longer commute to work, lower median household income, and lower rates of insurance coverage of children.

DETAILED DESCRIPTION:
The investigators will obtain HPV vaccine series completion data from the Indiana State Department of Health Immunization Information System (IIS) registry. The data will include all children 9 through 14 years of age who received the 1st dose of HPV vaccine during the 2017 and 2018 calendar years. A minimum of 18 months after 1st dose administration will be allowed for follow-up evidence of two-dose series completion. For comparison purposes, the investigators will also request Tdap, MenACWY, and HepA administration coverage. Tdap, MenACWY, and HepA vaccines are all required for middle-school-entry in the state of Indiana. The investigators already have data on missed opportunities for the 1st dose of HPV vaccine during the 2017 calendar year. Again, for comparison purposes, the investigators will request similar data for 2018. Tdap, MenACWY, and HepA administration rates will focus on children 11-14 years of age. County-level data will include measures of population density, primary health care providers per capita, mean household income, child insurance coverage, children living in poverty, length of work commute, participation in health screening behaviors, and other sociodemographic, health, and quality of life factors covered in CountyHealthRankings.Org.

the primary variable of interest is 2-dose series completion for HPV vaccination, measured via IIS data. All children and adolescents ages 9-14 years who received their first dose of vaccine during the 2017 and 2018 calendar years will be followed for series completion. For comparison purposes IIS data on Tdap, MenACWY, HepA, and HPV vaccine (missed opportunities for 1st dose) also will be derived from the IIS. Potential predictors of HPV vaccine series completion will be derived from CountyHealthRankings.Org. The County Health Rankings program is a collaborative effort of the Robert Wood Johnson Foundation and the University of Wisconsin Population Health Institute. Multiple health and sociodemographic indices measured at the county level are compiled and made publicly available on the website. As noted above, county-level measures derived from this program include population density, primary health care providers per capita, mean household income, child insurance coverage, children living in poverty, length of work commute, participation in health screening behaviors, and other sociodemographic, health, and quality of life factors covered in CountyHealthRankings.Org.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9 through 14 years of age in Indiana who received the first dose of HPV vaccine during the 2017 or 2018 calendar year.

Exclusion Criteria:

* Children younger than 9, as HPV vaccine is not licensed for children under 9 years of age
* Children older than 14 when they receive the first dose of vaccine

Ages: 9 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: All children with Indiana Immunization Information System (IIS) records who are 9 through 14 years of age and received their first dose of HPV vaccine during the 2017 or 2018 calendar years. All information on vaccination will be examined only at the county and state levels. No individual information will be used.
Sampling Method: Non-Probability Sample
Enrollment: 122152 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Percentage of children who complete the 2-dose HPV vaccine series | 2017-2020
  For those children aged 14 years and younger who received the first dose of HPV vaccine in 2017 or 2018 we will measure what percentage complete the second dose of vaccine during 18 months of follow-up.

SECONDARY OUTCOMES:
Percentage of children who receive other adolescent vaccines | 2017-2018
  Receipt of Tdap, MenACWY, and HepA vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No